CLINICAL TRIAL: NCT04339088
Title: Pilot Study to InVestigate the Efficacy and Safety of High Intensity Focused Ultrasound in PAtients With Varicose Veins in Singapore (VESPA)
Brief Title: High Intensity Focused Ultrasound in PAtients With Varicose Veins in Singapore
Acronym: VESPA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2933
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Varicose Veins; Venous Reflux; Chronic Venous Insufficiency
Keywords: Endovenous Ablation
MeSH Terms: conditions — Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIFU: Patients that have undergone high focused ultrasound treatment for varicose veins
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires to assess quality of life

SUMMARY:
The aim of the study is to evaluate the efficacy of non-invasive echotherapy for the treatment of varicose veins, within local population, using the Sonovein® device. The quality of life scores at baseline, 2 weeks, 3 months, 6 months and 12 months will be assessed using the EQ-50D, AVVQ and CIVIQ scores. Patient satisfaction at these time points will also be assessed.

DETAILED DESCRIPTION:
Sonovein® is a unique echotherapy solution, combining therapeutic ultrasound and ultrasound for monitoring. The high-intensity ultrasound beam is focused on the vein through a magnifying glass. As thermal energy is delivered, the thermocoagulation property of ultrasound energy affects the vein wall, causing shrinking and collapsing of the target vein. Thus creating a fibrotic seal and occluding the vessel. The treated vein is immediately closed after the procedure, and its diameter will continuously reduce over time, becoming a fibrotic chord. The treatment along the vein is steered automatically via a touch screen monitor. In-beam linear ultrasound probe allows visualisation of the vein in real-time and insures optimal accuracy. The study involves prospective data collection of 30 patients that will be undergoing HIFU as choice of treatment for their varicose veins / CVI. Questionnaires will be conducted at 5 timepoints - baseline before procedure, 2 weeks, 3 months, 6 months and 12 months. Subjects will be seen at outpatient clinic post-procedure. Besides questionnaires, physical examination and duplex ultrasound scan will be conducted at 2 weeks, 3 months, 6 months and 12 months to ensure occlusion of treated vein.

ELIGIBILITY:
Inclusion Criteria:

1. Age >21 years, able to understand the requirements of the study and provide informed consent.
2. C2 - C5 varicose veins / CVI
3. Symptomatic primary GSV, SSV or AASV incompetence, with reflux >0.5 seconds on colour duplex, including one or more of the following symptoms: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling.
4. Patients who has GSV, SSV or AASV diameters of 3mm to 12mm in the standing position.

Exclusion Criteria:

1. Current DVT or history of DVT
2. Recurrent varicose veins
3. Pregnant patients
4. Arterial disease (ABPI<0.8)
5. Sepsis
6. Patients who are unwilling to participate
7. Inability or unwillingness to complete questionnaires
8. Adverse reaction to sclerosant or cyanoacrylate
9. GSV, SSV or AASV severely tortuous
10. Life expectancy < 1 year
11. Active treatment for malignancy other than non-melanoma skin cancer
12. Current, regular use of systemic anticoagulation (e.g. warfarin, heparin)
13. Daily use of narcotic analgesia or NSAIDS to control pain associated with venous disease

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves prospective data collection of 30 patients that will be undergoing HIFU as a choice of treatment for their varicose veins / CVI.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical success at time of procedure | Immediately post-op
  Occlusion of treated vein post-procedure
Change in anatomy of treated vessel | 2 weeks, 3 months, 6 months, 12 months post-procedure
  Anatomical success as measured at each time-point using ultrasound to ensure occlusion of treated vein.

SECONDARY OUTCOMES:
Quality of life score using EQ-5D questionnaire | 2 weeks, 3 months, 6 months, 12 months post-procedure
  EQ5D is used to assess quality of life based on Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime.
Quality of Life Score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  CIVIQ is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging for 0 to 100 - the higher the value, the poorer the quality of life.
Quality of Life score using the Aberdeen Varicose Vein Questionnaire (AVVQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  To measure health status of varicose veins patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life
Clinical Change using Venous Clinical Severity Score (VCSS) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (mild), 2 (moderate), 3 (severe).
Pain Score | First 10 days post-procedure
  Using a numerical rating scale, which ranges from 0 (no pain) to 10 (severe pain)
Time taken to return to work and normal activities | 10 days post-operation
Occlusion rates | 2 weeks, 3 months, 6 months, 12 months post-procedure
  Duplex ultrasound performed at specific timepoints to ensure that treated vein is occluded
Patient satisfaction with treatment | 2 weeks, 3 months, 6 months, 12 months post-procedure
  A short survey to assess patient satisfaction and if there is any observed improvement in terms of appearance and symptoms post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapre General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Golledge J, Quigley FG. Pathogenesis of varicose veins. Eur J Vasc Endovasc Surg. 2003 Apr;25(4):319-24. doi: 10.1053/ejvs.2002.1843. PMID 12651169
- [Background] Callam MJ. Epidemiology of varicose veins. Br J Surg. 1994 Feb;81(2):167-73. doi: 10.1002/bjs.1800810204. PMID 8156326
- [Background] Tan KK, Nalachandran S, Chia KH. Endovenous laser treatment for varicose veins in Singapore: a single centre experience of 169 patients over two years. Singapore Med J. 2009 Jun;50(6):591-4. PMID 19551312
- [Background] Jawien A. The influence of environmental factors in chronic venous insufficiency. Angiology. 2003 Jul-Aug;54 Suppl 1:S19-31. doi: 10.1177/0003319703054001S04. PMID 12934754
- [Background] Navarro L, Min RJ, Bone C. Endovenous laser: a new minimally invasive method of treatment for varicose veins--preliminary observations using an 810 nm diode laser. Dermatol Surg. 2001 Feb;27(2):117-22. doi: 10.1046/j.1524-4725.2001.00134.x. PMID 11207682
- [Background] Law, Y., Chan, Y. C., Cheung, G. C. Y., Ting, A. C. W., Wong, A. C. C., & Cheng, S. W. K. (2016). Early single-centre comparative results on non-thermal ablation of symptomatic incompetent great saphenous veins (GSV): cyanoacrylate glue (VenaSeal) versus mechanicochemical ablation (ClariVein). Leipzig Interventional Course, LINC 2016.
- [Background] Teruya TH, Ballard JL. New approaches for the treatment of varicose veins. Surg Clin North Am. 2004 Oct;84(5):1397-417, viii-ix. doi: 10.1016/j.suc.2004.04.008. PMID 15364562
- [Background] Subramonia S, Lees T. Radiofrequency ablation vs conventional surgery for varicose veins - a comparison of treatment costs in a randomised trial. Eur J Vasc Endovasc Surg. 2010 Jan;39(1):104-11. doi: 10.1016/j.ejvs.2009.09.012. Epub 2009 Oct 29. PMID 19879166